CLINICAL TRIAL: NCT04689880
Title: A Prospective, Multicenter Study Evaluating the Safety and Performance of the NuVasive® XLIF Decade™ Plate System for the Treatment of Patients With Pathologic Conditions of the Thoracic and/or Lumbar Spine
Brief Title: XLIF Decade Plate System Study
Status: Completed | Type: Observational
Sponsor: NuVasive (Industry)
Responsible Party: Sponsor
Organization: Globus Medical Inc (Industry)
Other Study IDs: NUVA.DEC0820
Record Dates: First submitted 2020-12-28; First posted 2020-12-30 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Degenerative Disc Disease; Degenerative Spondylolisthesis; Degenerative Scoliosis
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: US Export: No

GROUPS / COHORTS (1):
- XLIF Decade Plate

SUMMARY:
The primary objective of this study is to evaluate the safety and performance of the NuVasive XLIF Decade Plate System as measured by patient-reported outcomes (PROs), radiographic outcomes, and reported complications.

DETAILED DESCRIPTION:
This study is a prospective, single-arm, multicenter study to evaluate the safety and performance of the XLIF Decade Plate in patients undergoing a thoracic and/or lumbar interbody fusion, at one or two levels, with supplemental fixation using a lateral plate. Consecutive patients at a given site who meet all eligibility requirements will be asked to consent to participate in the study. Eligible patients include those with degenerative conditions in the thoracic and/or lumbar spine that are amenable to surgical treatment and will be screened prior to study enrollment. Once enrolled in the study, subjects will undergo XLIF surgery with lateral plating using the Decade Plate. At least 75 subjects will be enrolled and will be followed for 24 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are ≥18 years of age at the time of consent
2. Planned interbody fusion surgery using the Decade Plate System in conjunction with an interbody implant to treat one or two levels in the thoracic and/or lumbar spine for

   1. degenerative disc disease
   2. spondylolisthesis
   3. scoliosis, kyphosis, lordosis
   4. spinal stenosis
   5. spondylolysis
   6. pseudoarthrosis or failed previous spine surgery
3. Able to undergo surgery based on physical exam, medical history, and surgeon judgment
4. Understands the conditions of enrollment, is willing to follow medical advice including postoperative activity restrictions per the surgeon's standard of care, and is willing to sign an informed consent form to participate in the study

Exclusion Criteria:

1. Use of posterior fixation for the scheduled surgery Note: Should the surgical plan change intraoperatively and posterior fixation is used in the case, the participant will be withdrawn from the study
2. Patient is involved in active litigation relating to the spine (worker's compensation claim is allowed if it is not contested)
3. Use of bone growth stimulators postoperatively
4. Active smoking within 6 weeks before surgery
5. Patient has known sensitivity to materials implanted
6. Systemic or local infection (latent or active) or signs of local inflammation
7. Patient has inadequate bone stock or quality, or a physical or medical condition that would prohibit beneficial surgical outcome based on surgeon judgment
8. Pregnant, or plans to become pregnant during the study
9. Patient is a prisoner
10. Patient is participating in another clinical study that would confound study data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Enrolled Population will include all subjects who meet the criteria for enrollment, specifically, those subjects who:
  * Satisfied the inclusion and exclusion criteria
  * Signed the informed consent
  * Underwent the surgical procedure, as defined in this protocol
  Subjects not meeting any of these criteria will not be considered enrolled in the study, and therefore not included in any study population or analysis.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Complication of interbody implant | 24 months
  Rate of device-related complications (i.e., safety) attributable to the use of the Decade Plate System
Radiographic fusion success | 24 months
  Proportion of subjects with apparent radiographic fusion (i.e., performance) of the index surgical level(s) at 24 months postoperative

SECONDARY OUTCOMES:
Percentage of subjects meeting minimal clinically important difference (MCID) as compared to baseline for back/leg pain measured by visual analog scale (VAS). | 24 months
  Back and leg pain measured using a visual analog scale (VAS) will be assessed to determine the percentage of subjects who meet MCID (1.2 points and 1.6 points respectively) where 0 is "No Pain" and 10 is "Unbearable Pain".
Percentage of subjects meeting minimal clinically important difference (MCID) as compared to baseline for disability measured by the Oswestry disability index. | 24 months
  Disability measured by the Oswestry disability index (ODI) will be assessed to determine the percentage of subjects who meet MCID (12.8 points) where a higher score on the ODI indicates a more severe disability.
Percentage of subjects meeting minimal clinically important difference (MCID) as compared to baseline measured by overall physical and mental health from PROMIS-10. | 24 months
  Overall physical and mental health measured by PROMIS-10 will be assessed to determine the percentage of subjects who meet MCID (5 points). PROMIS-10 scoring uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population.
Percentage of subjects meeting substantial clinical benefit (SCB) as compared to baseline for back/leg pain measured by visual analog scale (VAS). | 24 months
  Back and leg pain measured using a visual analog scale (VAS) will be assessed to determine the percentage of subjects who meet SCB (3.5 points or less, at least a 2.5 point improvement, or at least a 41.4% improvement) where 0 is "No Pain" and 10 is "Unbearable Pain".
Percentage of subjects meeting substantial clinical benefit (SCB) as compared to baseline for disability measured by the Oswestry disability index. | 24 months
  Disability measured by the Oswestry disability index (ODI) will be assessed to determine the percentage of subjects who meet SCB (at least 18.8 point improvement, at least a 36.8% improvement, or a disability value below 31.3) where a higher score on the ODI indicates a more severe disability.
Percentage of subjects meeting substantial clinical benefit (SCB) as compared to baseline measured by overall physical and mental health from PROMIS-10. | 24 months
  Overall physical and mental health measured by PROMIS-10 will be assessed to determine the percentage of subjects who meet MCID (7 points). PROMIS-10 scoring uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population.
Rate of complications attributable to the use of any additional NuVasive instruments, implants, or technologies. | 24 months
  Rate of complications attributable to the use of any additional NuVasive instruments, implants, or technologies

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Malone, MS, Study Director — NuVasive
Locations (1):
- Loma Linda University, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No